CLINICAL TRIAL: NCT03008369
Title: Phase II Trial of Lenvatinib in Metastatic or Advanced Pheochromocytoma and Paraganglioma
Brief Title: Lenvatinib in Treating Patients With Metastatic or Advanced Pheochromocytoma or Paraganglioma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1575; NCI-2016-02032 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1575 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Malignant Adrenal Gland Pheochromocytoma; Malignant Paraganglioma; Metastatic Adrenal Gland Pheochromocytoma
MeSH Terms: conditions — Paraganglioma, Extra-Adrenal; Pheochromocytoma | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenvatinib) (Experimental): Patients receive lenvatinib PO once daily on days 1-28. Courses repeat every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenvatinib; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenvatinib — Given PO
  Other Names: E7080; ER-203492-00; Multi-Kinase Inhibitor E7080
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies how well lenvatinib works in treating patients with pheochromocytoma or paraganglioma that has spread to other places in the body or cannot be removed by surgery. Lenvatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the anti-tumor activity of lenvatinib (overall response rate; [ORR]) in patients with metastatic or advanced unresectable pheochromocytomas and paragangliomas.

SECONDARY OBJECTIVES:

I. To determine progression-free survival (PFS). II. To determine overall survival (OS). III. To determine duration of tumor response. IV. To determine safety and tolerability of lenvatinib. V. To assess patient reported quality of life using EuroQol Five-Dimensional Five Level Scale Questionnaire (EQ-5D-5L) and Functional Assessment of Cancer Therapy-General (FACT-G).

TERTIARY OBJECTIVES:

I. For patients with secretory tumors, to examine changes in plasma metanephrine levels and urinary catecholamine and/or metanephrine levels.

II. For patients with secretory tumors, to examine whether lenvatinib-induced changes in plasma metanephrines and urinary catecholamine and/or metanephrine levels during the first cycle of treatment may be associated with objective tumor response.

III. To examine associations between tumor response and somatic mutational status in archived tumors, or germline mutational status (presence of SDHD, SDHB, RET, VHL, neurofibromatosis type-1).

OUTLINE:

Patients receive lenvatinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 or 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant secretory or non-secretory pheochromocytoma or paraganglioma that is unresectable and deemed inappropriate for alternative local regional therapeutic approaches
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Life expectancy > 24 weeks
* Absolute neutrophil count (ANC) >= 1500/mm^3
* White blood cell (WBC) count >= 3,000/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL (5.6 mmol/L); NOTE: transfusions are not allowed =< 7 days prior to registration
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (or total bilirubin =< 3.0 X ULN with direct bilirubin =< 1.5 X ULN in patients with well-documented Gilbert's Syndrome)
* Aspartate transaminase (AST/serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 X ULN
* Creatinine =< 1.5 x ULN
* Urine protein/creatinine ratio =< 1 OR 24-hour urine protein < 1.5 gram
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Blood pressure (BP) < 150 mmHg (systolic) and < 90 mmHg (diastolic); initiation or adjustment of BP medication is permitted prior to registration provided that the average of three BP readings at a visit prior to registration is < 150/90 mmHg; NOTE: all patients with secretory pheochromocytoma or paraganglioma are REQUIRED to: 1) be evaluated in consultation by a hypertension specialist with specific experience in the management of hypertension in the setting of catecholamine-secreting tumors (usually an endocrinologist, nephrologist, or a cardiologist), and in the setting of hormone-associated hypertension) receive alpha- and beta-adrenergic blockade for at least 7-14 days prior to initiation of lenvatinib; the hypertension specialist of record for each patient should be committed to closely following the patient during the clinical study with evaluation by said specialist required at cycle 1 and 2 and thereafter on an as needed basis
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Ability to complete questionnaire(s) by themselves or with assistance

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Chemotherapy/systemic therapy, radiotherapy, immunotherapy or surgery =< 21 days prior to registration or kinase inhibitor therapy =< 14 days prior to registration or failure to recover from toxicities (to grade 1 or below) from treatment; NOTE: concurrent therapy with octreotide is allowed providing that tumor progression on this therapy has been demonstrated; concurrent therapy with bisphosphonates (e.g. zoledronic acid) or denosumab is also allowed; NOTE: an unlimited number of prior chemotherapeutic or biologic therapies for malignant pheochromocytoma or paraganglioma is permitted; this includes prior anti-angiogenesis therapies such as tyrosine kinase inhibitors
* Active or uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent
* Current use of warfarin for any reason; NOTE: if patient can be safely transitioned to another anticoagulant, they may be eligible provided other criteria are satisfied
* Any of the following:

  * Correct QT (QTc) prolongation (defined as a QTc interval >= 500 msecs)
  * Left ventricular ejection fraction (LVEF) < institutional lower limits of normal (LLN)
  * Frequent ventricular ectopy
  * Evidence of ongoing myocardial ischemia
* Receiving any medications or substances with risk of torsades de pointes; NOTE: medications or substances with known risk of torsades de pointes are prohibited; consult pharmacist for review if needed
* Known active and/or untreated brain metastases
* Known severe allergic or other prohibitive reactions to other tyrosine kinase inhibitors (TKI)
* Prior treatment with lenvatinib
* Any of the following conditions:

  * Active peptic ulcer disease
  * Inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) or other gastrointestinal conditions which increase the risk of perforation
  * History of new abdominal fistula, gastrointestinal perforation or intra-abdominal abscess =< 84 days prior to registration; NOTE: enrollment of patients with chronic/canalized fistulous tracts (present for > 84 days) is allowed
  * Serious or non-healing wound, ulcer, or bone fracture
  * History of familial QTc prolongation syndrome
* Any of the following conditions =< 6 months prior to registration:

  * Cerebrovascular accident (CVA) or transient ischemic attack (TIA)
  * Serious or unstable cardiac arrhythmia
  * Admission for unstable angina or myocardial infarction
  * Cardiac angioplasty or stenting
  * Coronary artery bypass graft surgery
  * Pulmonary embolism, untreated deep venous thrombosis (DVT) or DVT which has been treated with therapeutic anticoagulation =< 30 days
  * Arterial thrombosis
  * Symptomatic peripheral vascular disease
* Other active malignancy =< 2 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer; NOTE: adjuvant anti-estrogen/hormonal therapy for breast cancer is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Chintakuntlawar, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Lenvatinib)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Lenvatinib): Patients receive lenvatinib PO once daily on days 1-28. Courses repeat every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity. Laboratory Biomarker Analysis: Correlative studies Lenvatinib: Given PO Quality-of-Life Assessment: Ancillary studies
Arm/Group | Treatment (Lenvatinib)
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 50 [44 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Tumor Response Rate
Description: Will be defined as 100% times the number of eligible patients who has started lenvatinib and whose objective tumor status was a complete response or partial response on 2 consecutive evaluations at least 4 weeks apart (using Response Evaluation Criteria in Solid Tumors version 1.1 criteria) divided by the number of eligible patients who has started lenvatinib. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Monthly, up to 17 months.
Measure: Number; unit: participants
Arm/Group | Treatment (Lenvatinib)
Number analyzed (Participants) | 3
participants | 1.0

2. Secondary Outcome: Duration of Tumor Response
Description: Will be estimated using the Kaplan-Meier method.
Time Frame: Every month until off treatment, at off treatment, every 3 months until PD, at PD, every 6 months after PD up to 17 months
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Lenvatinib)
Number analyzed (Participants) | 3
Months | 9.7 [9.7 to NA] — Upper limit not reached due to insufficient number of participants with events

3. Secondary Outcome: Patients Evaluable for Incidence of Adverse Events Assessed by Common Terminology Criteria for Adverse Events Version 4.0
Description: Adverse Events are fully reported in the adverse event section of the results. All adverse events will be graded. For each type of adverse event classified as either possibly, probably, or definitely related to study treatment, the proportion of patients experiencing a severe (grade 3 or higher) adverse event will be noted per cycle. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine adverse event patterns.
Time Frame: Monthly, up to 17 months.
Population: All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lenvatinib)
Number analyzed (Participants) | 3
Participants | 3

4. Secondary Outcome: Overall Survival Time
Description: Will be estimated using the Kaplan-Meier method.
Time Frame: as for outcome 2
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Lenvatinib)
Number analyzed (Participants) | 3
Months | NA [NA to NA] — Kaplan-Meier median, lower limit, and upper limit not reached due to insufficient number of participants with events.

5. Secondary Outcome: Progression-free Survival
Description: Will be estimated using the Kaplan-Meier method.
Time Frame: Every month until off treatment, at off treatment, every 3 months until PD, at PD or up to 17 months
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Lenvatinib)
Number analyzed (Participants) | 3
Months | 11.5 [5.5 to NA] — Upper limit not reached due to insufficient number of participants with events

6. Secondary Outcome: Quality of Life Assessed by EQ-5D and FACT-G
Description: Descriptive statistics, and scatter plots will form the basis of presentation of these data both overall and by other outcomes (toxicity, response and survival measures). Correlations between the quality of life outcomes and other outcome measures will be carried out by standard parametric and nonparametric tests (e.g. Pearson's and Spearman's rho). Comparison between continuous variables will be made with Wilcoxon rank sum tests, Fisher's exact tests will be used to determine differences between categorical variables, and Log-rank test will be used to test differences between time-to-event ou
Time Frame: 5 years
Population: No patients made it to the QoL timepoint or submitted QoL data after treatment.
Arm/Group | Treatment (Lenvatinib)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Changes in Urinary Catecholamine and Metanephrine Levels
Description: Wilcoxon rank sum tests will be used to examine whether fold changes in a given biomarker during the first cycle of treatment differs between whose tumor responded to treatment and those whose tumor did not. Time series plots will be constructed.
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Germline Mutational Status in Peripheral Blood Mononuclear Cells
Description: Will examine associations between tumor response and somatic mutational status in archived tumors, or germline mutational status in patient's peripheral blood mononuclear cells, (presence of SDHD, SDHB, RET, VHL, neurofibromatosis type-1).
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Somatic Mutational Status in Peripheral Blood Mononuclear Cells
Description: as for outcome 8
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Monthly, up to 17 months.
Description: Incidence of Adverse Events Assessed by Common Terminology Criteria for Adverse Events Version 4.0
Arm/Group | Treatment (Lenvatinib)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenvatinib) (N=3)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenvatinib) (N=3)
Hyperthyroidism (Endocrine disorders) | 2 (4)
Hypothyroidism (Endocrine disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (12)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (11)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (19)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (4)
Proteinuria (Renal and urinary disorders) | 3 (15)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (4)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 1 (4)
Hypertension (Vascular disorders) | 2 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT03008369/Prot_SAP_000.pdf